CLINICAL TRIAL: NCT03950726
Title: Minimally Invasive Open Technique for Ileo-colic Resection in Complex Cases of Terminal Ileum Crohn's Disease. Case Series.
Brief Title: Ileocolic Resection for Complex Crohn's Disease
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, simone sibio, associate professor, University of Roma La Sapienza
Other Study IDs: Chirurgia Mini-invasiva PTV
Record Dates: First submitted 2019-05-07; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Crohn Disease of Ileum
Keywords: Crohn Disease; Ileocolic resection; Appendectomy; Single-port incision; McBurney; Laparoscopy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: patients with complex crohn's disease who had a previous open appendectomy through a mc burney incision scheduled for ileo-colic resection through the same incision
  Interventions: Procedure: ileocolic resection
- Control Group: patients with complex crohn's disease who had a previous open appendectomy through a mc burney incision scheduled for ileo-colic resection who underwent standard laparoscopic resection
  Interventions: Procedure: ileocolic resection

INTERVENTIONS:
Procedure: ileocolic resection — Ileocolic resection through McBurney incision

SUMMARY:
Laparoscopic ileocolic resection is the preferred surgical approach for patients with ileocecal Crohn's disease (CD). Objective of this study was to evaluate the efficacy of a minimally invasive gas-less ileocolic resection in complex cases of CD through a Mc Burney incision, in patients who already had a previous appendectomy.

DETAILED DESCRIPTION:
From January 2016 to December 2017, all consecutive CD patients with primary or recurrent complex disease referred for IC resection were evaluated for the study purpose.Complex disease patients presenting McBurney incision for a previous open appendectomy were included in the group of study. This group was compared with a control group of CD patients with the same clinical characteristics of ileocolic disease who underwent standard laparoscopic IC resection, pooled out from the database of IC resections for CD of the Minimally Invasive and Gastrointestinal Surgery Unit of Tor Vergata Hospital, Rome, Italy. Data on demographics, BMI, type and behavior of CD, presence of disease apart from ileocecal site, previous surgery, recurrence, current medical treatment, thickening of the mesentery, preoperative imaging results (MR enterography or small intestine contrast ultrasound), operative time, blood loss, conversion to laparoscopy and conversion to open rates, complications, adherence rate to ERAS protocols and length of hospital stay were collected for the study purpose.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed Crohn's disease
* previous appendectomy trough a mcburney incision

Exclusion Criteria:

* patients with major comorbidities
* age>75
* previous midline laparotomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with complex terminal ileum Crohn's disease candidate for ileocolic resection who underwent to previous open appendectomy.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-05-04 (Actual)

PRIMARY OUTCOMES:
Mean operative time | 75-156 minutes
  duration of surgical procedure
Mean blood loss during surgical procedure | 2 hours
  blood loss from the beginning to the end of the procedure
Mean post-operative hospital stay | 3-7 days
  time from day of surgery to discharge

SECONDARY OUTCOMES:
post-operative complications | 30 days
  complications according to Clavien Dindo classification